CLINICAL TRIAL: NCT01388088
Title: Effect of Amiloride and Spironolactone on Renophysiological and Cardiovascular Variables in Patients With Essential Hypertension in a Doublle-blinded Randomised Placebo-controlled, Cross-over Study.
Brief Title: The Effect of Amiloride and Spironolactone in Patients With Hypertension
Acronym: hass
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erling Bjerregaard Pedersen (Other)
Responsible Party: Sponsor-Investigator, Erling Bjerregaard Pedersen, Proffesor, Regional Hospital Holstebro
Organization: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MED.RES.HOS.2010.02.SKM
Record Dates: First submitted 2010-05-19; First posted 2011-07-06 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Hypertension
Keywords: Hypertension; Potassium; Blood-pressure
MeSH Terms: conditions — Hypertension | interventions — Spironolactone; Amiloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Spironolactone (Active Comparator): Increases the level of potassium
  Interventions: Drug: Spironolactone
- Amiloride (Active Comparator): Increases the level of potassium
  Interventions: Drug: Amiloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — 25 mg twice a day
  Arms: Spironolactone
Drug: Amiloride — 5 mg twice a day
  Arms: Amiloride
Drug: Placebo — twice a day
  Arms: Placebo

SUMMARY:
The investigators wish to investigate the potential effects of potassium. In this study we will examine patients with hypertension and increase their potassium-levels using Amiloride and Spironolactone.

The investigators will examine the changes in the cardiovascular system using a Sphygmocor-scanner.

DETAILED DESCRIPTION:
Purpose of the study is to examine the effect of amilorid and spironolacton on

1. Renal function (GFR, u-AQP2, u-ENaCβ, u-cAMP, u-PGE2, CH20, FENa, FEK),
2. Pulsewavevelocity, augmentation index and centralt bloodpressure,
3. Vasoactive hormones (PRC, AngII, Aldo, AVP, ANP, BNP and Endot), and
4. Ambulatory blood pressure

ELIGIBILITY:
Inclusion Criteria:

* Hypertension
* Age 45-70
* BMI: 18,5-30

Exclusion Criteria:

* Other diseases
* Drug or alcohol abuse
* Abnormal findings in the screening procedure

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 2 years
  24 hours blood pressure measurements

SECONDARY OUTCOMES:
Pulse wave velocity | 2 years
  We will investigate the changes in cardiovascular variables using a Sphygmocor scanner.

CONTACTS AND LOCATIONS:
Overall Officials: Solveig K Matthesen, Cand.Med, Principal Investigator — Medical Research Department
Locations (1):
- Department of Medical Research, Holstebro, Denmark